CLINICAL TRIAL: NCT00516906
Title: Clinical Performance of a Chlorhexidine Antimicrobial Dressing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: University of Nebraska (Other); 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-010691
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Results first posted 2012-02-23 (Estimated); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Catheterization
MeSH Terms: interventions — chlorhexidine gluconate; DAT protocol 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transparent Adhesive Dressing (Placebo Comparator): Standard of Care Non-Antimicrobial Transparent Adhesive Dressing
  Interventions: Drug: Transparent Adhesive Dressing
- CHG antimicrobial transparent dressing (Experimental): Chlorhexidine gluconate antimicrobial transparent adhesive dressing
  Interventions: Drug: Chlorhexidine gluconate

INTERVENTIONS:
Drug: Chlorhexidine gluconate — 2% Chlorhexidine Transparent Dressing applied as needed up to 7 days of wear
  Other Names: 3M(TM) Tegaderm(TM) CHG Dressing
  Arms: CHG antimicrobial transparent dressing
Drug: Transparent Adhesive Dressing — Standard of Care Non-antimicrobial Transparent Adhesive Dressing applied as needed for up to 7 days of wear
  Other Names: TAD, Polyurethane Dressing, Transparent Membrane Dressing
  Arms: Transparent Adhesive Dressing

SUMMARY:
Evaluate the clinical performance of a new IV Dressing in Comparison to a standard IV Dressing

DETAILED DESCRIPTION:
Prospective, controlled, randomized, clinical trial comparing the 3M™ TegadermTM CHG (Chlorhexidine Gluconate) IV Securement Dressing (3M Healthcare, St Paul, MN) to a standard transparent dressing.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females over 18 years of age
* Patients with an existing, or newly inserted, central venous catheter
* Patients who require the catheter for at least 3 days

Exclusion Criteria:

* Sensitivity to chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Rupp, M.D., Principal Investigator — Nebraska Medical Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included adult males and female patients with an existing, or newly inserted, catheter that was to remain in place for at least 3 days, who were willing to participate in the study, and who would provide informed consent and sign a consent form. First patient enrolled 10 October 2007. Last patient enrolled 20 December 2007
Pre-assignment Details: No Wash out. No run-in
Groups:
- Placebo Comparator: A: Standard of Care Transparent Adhesive Dressing
Period: Overall Study
Arm/Group | Placebo Comparator: A | CHG Antimicrobial Transparent Dressing
Started | 36 | 32 (33 patients were randomized but one patient was discharged prior to treatment.)
Completed | 30 (Thirty patients were required to complete. Patients not completing were replaced.) | 30 (Thirty patients were required to complete. Patients not completing were replaced.)
Not Completed | 6 | 2
Not completed — Final Dressing Removal Data not captured | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: A | CHG Antimicrobial Transparent Dressing | Total
Number analyzed (Participants) | 36 | 32 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 45
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (15.1) | 53.4 (18.5) | 56.0 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 36 | 32 | 68

OUTCOME MEASURES:

1. Primary Outcome: Clinician Overall Satisfaction With Catheter Securement
Description: Clinician Overall Satisfaction with Catheter Securement Five Point Scale: 1 = Very Good, 5= Very Poor
Time Frame: Daily up to 7 Days (average 3-7 days of wear)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Comparator: A | CHG Antimicrobial Transparent Dressing
Number analyzed (Participants) | 30 | 30
Units on a scale | 2.27 (0.78) | 1.63 (1.63)

2. Secondary Outcome: Clinician Overall Satisfaction With Dressing
Description: Clinician Overall Satisfaction with Dressing Five point scale: 1= Very Good, 5= Very poor
Time Frame: Daily up to 7 Days (average 3-7 days of wear)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Comparator: A | CHG Antimicrobial Transparent Dressing
Number analyzed (Participants) | 30 | 30
Units on a scale | 2.20 (0.81) | 1.63 (0.61)

3. Secondary Outcome: Rating of Skin Condition
Description: Ratings of skin condition for erythema on a 0 to 3 scale (0 = None, 1=Mild, 2=Moderate, 3=Severe)
Time Frame: Daily up to 7 Days (average 3-7 days of wear)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Comparator: A | CHG Antimicrobial Transparent Dressing
Number analyzed (Participants) | 30 | 30
Units on a scale | 0.1 (0.29) | 0.2 (0.33)

ADVERSE EVENTS:
Time Frame: The study ran 3 months (10 October 2008- 20 December 2008) The maximum length of exposure of each patient to the dressings was 7.1 days.
Description: The insertion site was evaluated each day by study personnel and patients were asked about their well being
Arm/Group | Placebo Comparator: A | CHG Antimicrobial Transparent Dressing
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/30
Other Adverse Events (participants affected / at risk) | 2/30 | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: A (N=30) | CHG Antimicrobial Transparent Dressing (N=30)
Death due to underlying Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: A (N=30) | CHG Antimicrobial Transparent Dressing (N=30)
Elevated Temperature (General disorders) | 1 (1) | 1 (1)
Elevated WBC, No fever, culture negative (Infections and infestations) | 1 (1) | 0 (0)
Intermittent confusion existing prior to start (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial evaluated the dressing for it's securement and ease of use adaption into healthcare practices compared to a standard transparent dressing. The sample size was too small to evaluate any effect on Catheter Related-Bloodstream Infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No